CLINICAL TRIAL: NCT06291129
Title: Assessment of Oral Hygiene, Gingival Health, and Malocclusion Among Type 1 Diabetic Children and Adolescents: an Original Article
Brief Title: Gingival Health and Malocclusion Among Type 1 Diabetic Children and Adolescents
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Principal Investigator, Gabriela Alessandra da Cruz Galhardo Camargo, PhD, Universidade Federal Fluminense
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CAAE: 61347422.4.0000.5626
Record Dates: First submitted 2023-11-20; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Gingivitis; Periodontal Diseases; Diabetes; Diabetes Mellitus, Type 1; Malocclusion; Malocclusion in Children
MeSH Terms: conditions — Gingivitis; Periodontal Diseases; Diabetes Mellitus; Diabetes Mellitus, Type 1; Malocclusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hematological and Periodontal Parameters (Other): Hematological parameters were recorded - fasting blood glucose and glycosylated hemoglobin - to confirm the allocation of each participant between the groups: diabetic (DM) and control (NDM). The clinical periodontal parameters, including plaque index (PI) and bleeding on probing (GI) full mouth (Ainamo & Bay 1975), and plaque index (PI), probing depth of pocket (PPD), gingival recession (GR) and clinical attachment level (CAL). Gingival biotype clinical parameters were evaluated by three aspects: Gingival transparency to probing, Height of keratinized mucosa and Gingival thickness on permanent incisors and molars. For the periodontal parameters' examination, a periodontal probe PCP15 (PCP-UNC15, Hu-Friedy, Chicago, IL) was used, excluding third molars and erupting teeth. The intraexaminer agreement of the categorical variables (CAL) using the kappa calculation was 7.64, at the tooth level.
  Interventions: Procedure: Periodontal therapy
- Orthodontic Parameters (No Intervention): The clinical orthodontic parameters were recorded by the Angle's Classification, witch evaluated occlusion of right and left canines and molars, and the Dental Aesthetic Index (DAI) that evaluates the prevalence of malocclusions, its severity and the need for treatment. DAI aspects evaluated were: upper teeth loss, lower teeth loss, crowding, spacing, diastema, maxillary misalignment, mandibular misalignment, anterior maxillary overjet, anterior mandibular overjet, anterior open bite, molar relationship.

INTERVENTIONS:
Procedure: Periodontal therapy — Supragingival scaling sessions were performed with ultrasonic scalers (Dabi Atlante, Rio de Janeiro, RJ, Brazil) to remove all calculus and biofilms, in addition to oral hygiene guidelines, including brushing technique and interdental cleaning with dental floss.
  Arms: Hematological and Periodontal Parameters

SUMMARY:
Introduction: This study aims to evaluate the gingivitis, periodontal profile and malocclusion in children and adolescents with diabetes. Methods: The sample consisted of 36 children, who were distributed into two groups: DM; n=18 and NDM; n=18. Periodontal parameters considered were plaque Index (PI), gingival Index (GI), probing depth of pocket (PPD), gingival recession (GR) and clinical attachment level (CAL). Gingival biotype clinical parameters: Gingival transparency to probing, Height of keratinized mucosa and Gingival thickness on permanent incisors and molars. Malocclusion were evaluated by the Dental Aesthetic Index (DAI) and the Angle's Classification. The statistical analyses were Shapiro Wilk test and T test.

DETAILED DESCRIPTION:
Introduction: This study aims to evaluate the gingivitis, periodontal profile and malocclusion in children and adolescents with diabetes. Methods: The sample consisted of 36 children (age 8 to 18 years old), who were distributed into two groups: patients with type 1 diabetes (DM; n=18) and control patients without diabetes (NDM; n=18). Periodontal parameters considered were plaque Index (PI), gingival Index (GI), probing depth of pocket (PPD), gingival recession (GR) and clinical attachment level (CAL). Gingival biotype clinical parameters were evaluated by three aspects: Gingival transparency to probing, Height of keratinized mucosa and Gingival thickness on permanent incisors and molars. Malocclusion, its prevalence, severity and need of treatment were evaluated by the Dental Aesthetic Index (DAI) and the Angle's Classification. The statistical analyses were Shapiro Wilk test and T test.

ELIGIBILITY:
Inclusion Criteria:

- child or adolescent with the age between 8 and 18 years old

Exclusion Criteria:

* child or adolescent who had an active or inactive caries lesion, on the buccal surface, in the cervical region of the elements to be analyzed;
* participants with probing depth greater than or equal to 4 mm, which is characterized as periodontitis;
* the patient who is undergoing orthodontic treatment, with fixed appliance;
* smokers;
* pregnant women, nursing mothers.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-10-30 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Bleeding on probing | Twenty-one days
  Bleeding levels on probing below 10% of the periodontal sites evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela C Cruz, PhD, Principal Investigator — Universidade Federal Fluminense
Locations (1):
- Universidade Federal Fluminense, Nova Friburgo, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No